CLINICAL TRIAL: NCT02022813
Title: Impact of Supplemental Parenteral Nutrition (SPN) on Energy Balance, and Infection Rate in Intensive Care Patients: Underlying Metabolic, Inflammatory and Immune Mechanisms.
Brief Title: Impact of Supplemental Parenteral Nutrition in ICU Patients on Metabolic, Inflammatory and Immune Responses
Acronym: SPN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Mette M Berger, Prof, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CE 371-13
Record Dates: First submitted 2013-11-25; First posted 2013-12-30 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2016-02

CONDITIONS: Critical Illness
Keywords: Energy requirements, Glucose turnover, Protein turnover
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral nutrition only (No Intervention): Enteral nutrition to be progressed as soon as possible to energy target measured on day 3, and verified on day 4, using the usual facilitators (prokinetics)
- Supplemental parenteral nutrition (Experimental): Addition of supplemental parenteral nutrition to complete the gap between energy delivered by enteral feeding and energy target measured on day 4.
  Aim: 100% of this target, and not exceeding it, no catch up for energy deficit accumulated before day 4.
  Interventions: Dietary Supplement: Supplemental parenteral nutrition (SPN)

INTERVENTIONS:
Dietary Supplement: Supplemental parenteral nutrition (SPN) — The amount of energy delivered by SPN will depend on the indirect calorimetry measurement and actual enteral feed delivery. SPN will be reduced with progressing EN
  Other Names: Standard industrial PN solutions
  Arms: Supplemental parenteral nutrition

SUMMARY:
Having previously demonstrated that supplemental parenteral nutrition to complete an insufficient enteral nutrition (EN) between D4 and D8 improves outcome after critical illness, by reducing infectious complications, the present trial aims at investigating the underlying carbohydrate and protein metabolism changes, as well as the immune and inflammatory modulations associated with this improvement.

DETAILED DESCRIPTION:
Enrollment on day 3 of critically ill patients, without contraindication to EN, not achieving 60% of the ICU per protocol energy target.

Intervention: Randomization to either continued pure EN, or from day 4 to supplemental PN to complete EN at target validated by indirect calorimetry.

Measurements: Indirect calorimetry on Days 3, 4, 9 (twice). Primary endpoints = glucose and leucine metabolism On days 4 and 9-10: isotopic investigation of glucose metabolism, and immune and inflammatory responses// Day 9-10: isotopic investigation of protein (leucine) metabolism Secondary endpoints: Insulin requirements, area under the curve (AUC) of blood Glucose, infections after day 9, overall complications, length of mechanical ventilation, of ICU and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* estimated duration of ICU stay > 5 days,
* estimated survival > 7 days,
* absence of contraindication to EN
* need for mechanical ventilation
* informed consent obtained from patients, close relative, or referring physician

Exclusion Criteria:

* refusal of the patient or of the next of kin
* age < 18 years
* non-functional digestive tract (short bowel, persistent ileus, proximal intestinal fistula high rate > 1.5 litres/day)
* already receiving PN before Day 3
* absence of a central venous catheter
* women who are pregnant (pregnancy test).
* Admission after cardiac arrest, or severe brain injury

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Glucose and Leucine turnover | 10 days
  On D04:Infusion after priming of 6.6 2H2 glucose and NaH13CO3 On Day 09-10: Infusion after priming of NaH13CO3 and of L-[1-13C]-Leucine + repeat of the glucose sequence

SECONDARY OUTCOMES:
Immune and inflammatory impact of optimized target feeding | 10 days
  lymphocyte phenotypes: lymphocyte subpopulations (frequency), level of activation (CD69), memory markers, effectors, regulators
  * Cluster differentiation CD4, CD8, and natural killer (NK) phenotypes
  * Cell inflammatory response (WBA and PBMC) on D4 and D10±1: IL-2, TNF-α, interleukine-6 (IL-6), IL-1, TGF, IL-10, in culture for 24 to 48h ex vivo and post stimulation by memory mix and mitogens.
  * Serological inflammatory response (WBA and PBMC) on D4 and D10+1: TNF-α , IL-6, C-reactive protein (CRP): ex vivo with ELISA Nosocomial infections after day 8

OTHER OUTCOMES:
Global outcome | 28 days / 90 days
  Overall complications and organ failures, length of mechanical ventilation, length of ICU and hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Berger, MD PhD, Principal Investigator — CHUV, Lausanne
Locations (2):
- Switzerland (2):
  - Nutrition Unit, Geneva University Hospital, Geneva, Canton of Geneva
  - Service of Adult Intensive Care - CHUV, Lausanne, Canton of Vaud

REFERENCES:
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Derived] Berger MM, Pantet O, Jacquelin-Ravel N, Charriere M, Schmidt S, Becce F, Audran R, Spertini F, Tappy L, Pichard C. Supplemental parenteral nutrition improves immunity with unchanged carbohydrate and protein metabolism in critically ill patients: The SPN2 randomized tracer study. Clin Nutr. 2019 Oct;38(5):2408-2416. doi: 10.1016/j.clnu.2018.10.023. Epub 2018 Nov 5. PMID 30448193